CLINICAL TRIAL: NCT04846283
Title: Drainage Fluid Biomarkers And Anastomotic Leakage In Colorectal Surgery. A Monocentric Prospective Observational Study
Acronym: ALbiomarkers
Status: Completed | Type: Observational
Sponsor: University of Palermo (Other)
Responsible Party: Principal Investigator, Prof. Antonino Agrusa, Associate professor, University of Palermo
Other Study IDs: ANASTOMOTICLEAKAGE 01_2021
Record Dates: First submitted 2021-04-09; First posted 2021-04-15 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Anastomotic Leakage
Keywords: Anastomotic leakage; Colorectal surgery; Biomarkers
MeSH Terms: conditions — Anastomotic Leak | interventions — Elective Surgical Procedures

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Biomarker-group: We considered for the study all patients aged >16 y undergoing elective or emergency colorectal surgery for cancer, diverticular disease, inflammatory bowel-disease or reversal of Hartmann's procedure. Both patients undergoing open and minimally invasive surgery were considered eligible.
  Interventions: Procedure: Elective or emergency colorectal surgery for cancer, diverticular disease, inflammatory bowel-disease or reversal of Hartmann's procedure

INTERVENTIONS:
Procedure: Elective or emergency colorectal surgery for cancer, diverticular disease, inflammatory bowel-disease or reversal of Hartmann's procedure — We considered all the procedures that required an intestinal anastomosis in colo-rectal surgery

SUMMARY:
Anastomotic leakage (AL) is one of the most feared intra-abdominal septic complications (IASC) after colorectal surgery. It is defined as the leak of intestinal content due to an anastomotic dehiscence. Incidence ranges from 2% to 20%. AL is usually associated to systemic inflammatory response, even if in some cases the presentation may be subclinical. Therefore, AL is suspected in patients with a strong inflammatory response and can be confirmed by imaging with contrast enhanced computed tomography (CT) scan or water-soluble contrast studies. Nevertheless, imaging has varying sensitivity and specificity and is usually performed once the patient has a clinical evidence, thus potentially delaying the correct timing for surgery. Despite several studies about this topic and the plenty of known risk factors as mentioned above, AL is still not easy to predict. Different tools other than imaging have been studied in order to make diagnosis of AL at an early stage, as the measurement of some biomarkers of inflammation in serum and in drainage fluid.

Biomarkers as white cell blood count (WBC), C-reactive protein (CRP), cytokines (e.g. TNFa, IL-6, IL-1b), markers of ischemia (e.g. lactate) and procalcitonin (PCT) have been used for an early detection of AL and other intra-abdominal septic complications. The primary aim of our study was to assess the role of drainage fluid CRP and lactate-dehydrogenase (LDH) in the early detection of anastomotic leakage.

ELIGIBILITY:
Inclusion Criteria:

* patients aged >16 y undergoing elective or emergency colorectal surgery for cancer
* patients aged >16 y undergoing elective or emergency colorectal surgery for diverticular disease
* patients aged >16 y undergoing elective or emergency colorectal surgery for inflammatory bowel-disease
* patients aged >16 y undergoing elective or emergency colorectal surgery for reversal of Hartmann's procedure.

Exclusion Criteria:

* patients aged < 16 y undergoing colorectal surgery;
* patients undergoing Hartman's procedure

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients undergoing elective or emergency colorectal surgery for cancer, diverticular disease, inflammatory bowel-disease or reversal of Hartmann's procedure
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2020-04-01 (Actual); Study Completion 2020-04-01 (Actual)

PRIMARY OUTCOMES:
Measurement of drainage fluid CRP and LDH on postoperative day 3 | Postoperative day 3
  Our primary endpoint was to assess the role of drainage fluid CRP and LDH on postoperative day 3.

OTHER OUTCOMES:
Measurement of drainage fluid pH | Postoperative day 3
  Drainage fluid pH measurements were recorded on postoperative day 3 before drain removal.

CONTACTS AND LOCATIONS:
Overall Officials: Antonino Agrusa, Professor, Principal Investigator — University of Palermo - Italy
Locations (1):
- A.U.O. Azienda Ospedaliera Universitaria Policlinico "P. Giaccone" Palermo - University of Palermo, Palermo, Italy - Sicily, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smith SR, Pockney P, Holmes R, Doig F, Attia J, Holliday E, Carroll R, Draganic B. Biomarkers and anastomotic leakage in colorectal surgery: C-reactive protein trajectory is the gold standard. ANZ J Surg. 2018 May;88(5):440-444. doi: 10.1111/ans.13937. Epub 2017 Mar 17. PMID 28304142
- [Background] Molinari E, Giuliani T, Andrianello S, Talamini A, Tollini F, Tedesco P, Pirani P, Panzeri F, Sandrini R, Remo A, Laterza E. Drain fluid's pH predicts anastomotic leak in colorectal surgery: results of a prospective analysis of 173 patients. Minerva Chir. 2020 Feb;75(1):30-36. doi: 10.23736/S0026-4733.19.08018-0. Epub 2019 Sep 30. PMID 31580043
- [Background] Straatman J, Cuesta MA, Tuynman JB, Veenhof AAFA, Bemelman WA, van der Peet DL. C-reactive protein in predicting major postoperative complications are there differences in open and minimally invasive colorectal surgery? Substudy from a randomized clinical trial. Surg Endosc. 2018 Jun;32(6):2877-2885. doi: 10.1007/s00464-017-5996-9. Epub 2017 Dec 27. PMID 29282574
- [Background] Pedrazzani C, Moro M, Mantovani G, Lazzarini E, Conci S, Ruzzenente A, Lippi G, Guglielmi A. C-reactive protein as early predictor of complications after minimally invasive colorectal resection. J Surg Res. 2017 Apr;210:261-268. doi: 10.1016/j.jss.2016.11.047. Epub 2016 Dec 5. PMID 28457337
- [Background] Cabellos Olivares M, Labalde Martinez M, Torralba M, Rodriguez Fraile JR, Atance Martinez JC. C-reactive protein as a marker of the surgical stress reduction within an ERAS protocol (Enhanced Recovery After Surgery) in colorectal surgery: A prospective cohort study. J Surg Oncol. 2018 Mar;117(4):717-724. doi: 10.1002/jso.24909. Epub 2018 Jan 22. PMID 29355975
- [Background] Wright EC, Connolly P, Vella M, Moug S. Peritoneal fluid biomarkers in the detection of colorectal anastomotic leaks: a systematic review. Int J Colorectal Dis. 2017 Jul;32(7):935-945. doi: 10.1007/s00384-017-2799-3. Epub 2017 Apr 12. PMID 28401350
- [Background] Walker PA, Kunjuraman B, Bartolo DCC. Neutrophil-to-lymphocyte ratio predicts anastomotic dehiscence. ANZ J Surg. 2018 Jan 27. doi: 10.1111/ans.14369. Online ahead of print. PMID 29377500
- [Background] Reynolds IS, Boland MR, Reilly F, Deasy A, Majeed MH, Deasy J, Burke JP, McNamara DA. C-reactive protein as a predictor of anastomotic leak in the first week after anterior resection for rectal cancer. Colorectal Dis. 2017 Sep;19(9):812-818. doi: 10.1111/codi.13649. PMID 28273409
- [Derived] Agnello L, Buscemi S, Di Buono G, Vidali M, Lo Sasso B, Agrusa A, Ciaccio M. Drainage fluid LDH and neutrophil to lymphocyte ratio as biomarkers for early detecting anastomotic leakage in patients undergoing colorectal surgery. Clin Chem Lab Med. 2023 Nov 22;62(5):967-978. doi: 10.1515/cclm-2023-1164. Print 2024 Apr 25. PMID 37988156